CLINICAL TRIAL: NCT03239405
Title: Comparing the Cost Savings Potential of Orogastric Tubes in Laparoscopic Sleeve Gastrectomy
Acronym: VS1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boehringer Labs LLC (Industry)
Collaborators: Rochester General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VIS-1
Record Dates: First submitted 2017-07-27; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-07

CONDITIONS: Surgical Procedure, Unspecified
Keywords: laparoscopic; sleeve; gastrectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- SCS: Treated via suction callibrated system
  Interventions: Device: Suction callibrated system
- Bougie: Treated with multiple tubes & bougie

INTERVENTIONS:
Device: Suction callibrated system — One-step suction callibrated SG system
  Other Names: Visigi 3D
  Groups: SCS

SUMMARY:
Comparing the operation times and staple loads used between the use of multiple tubes and a bougie versus a one-step suction callibrated system in laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
In this study we are comparing the cost/savings of using a bougie with a one-step suction callibrated system in laparoscopic sleeve gastrectomy. We will be looking at OR time and staple usage. This study is not affecting the treatment of the patients in any way. The surgeons would be using the devices regardless of the study. We are simply looking at procedure information after the fact.

ELIGIBILITY:
Inclusion Criteria:

* Patient and surgeon have both agreed that a sleeve gastrectomy is a procedure that they want performed.

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals already receiving a laparoscopic sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Staples Used | 4 hours for the end of surgery
  Number of staple loads needed to close stomach
Operation time | 4 hours for the end of surgery
  Total operation time

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester General, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
Results will be published